CLINICAL TRIAL: NCT06476704
Title: Phase 2 Study of Preoperative RAdiation Therapy With Concomitant Liposomal Transcrocetin (L-TC) in Soft tISsue Sarcomas
Brief Title: Study of Preoperative RAdiation Therapy With Concomitant Liposomal Transcrocetin (L-TC) in Soft tISsue Sarcomas
Acronym: PRACTISS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: LEAF4Life, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-016; 2024-515668-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Sarcoma
Keywords: hypofractionated radiotherapy; soft tissue sarcoma; hypoxia; liposomal transcrocetin; neo-adjuvant
MeSH Terms: conditions — Sarcoma; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hypofractionated radiotherapy + Liposomal Transcorcetin (L-TC) (Experimental): L-TC as an IV infusion over 90 minutes at a fixed dose of 300 mg daily before each HFRT fraction, for a total of 5 days corresponding to the planned five daily HFRT fractions. The intravenous infusion should begin 2 hours before each HFRT fraction. Radiotherapy is scheduled to coincide with the plasma peak, which occurs approximately 2 hours after the start of the infusion. + HFRT treatment will be administered in control group as 30 Gy in 5 fractions of 6 Gy. 1 fraction per day, 5 days per week.
  Interventions: Drug: Administration of L-TC
- Hypofractionated radiotherapy alone (Active Comparator): HFRT treatment will be administered in control group as 30 Gy in 5 fractions of 6 Gy. 1 fraction per day, 5 days per week.
  Interventions: Radiation: HFRT alone

INTERVENTIONS:
Drug: Administration of L-TC — Administration of L-TC (300 mg) as an IV perfusion, daily before each radiotion session
  Arms: Hypofractionated radiotherapy + Liposomal Transcorcetin (L-TC)
Radiation: HFRT alone — HFRT : 30 Gy in 5 fractions of 6 Gy.
  1 fraction per day, 5 days per week.
  Arms: Hypofractionated radiotherapy alone

SUMMARY:
This is phase II randomized, multicenter study of treatment with L-TC and preoperative HFRT in patients who were aged 18 years or older with documented localised or locally advanced soft-tissue sarcoma of the extremity.

Eligible patients will be randomly assigned 2:1 to receive a preoperative HFRT alone (Arm A) or L-TC with preoperative HFRT (Arm B).

DETAILED DESCRIPTION:
This is a non-comparative phase II trial (comparison is made regarding a reference, not 2 between 2 proportions). Considering the wide confidence interval retrieved in literature regarding pCR value with HFRT, pCR value used in the sample size calculation and taken from the literature must be included in the 95% CI of the pCR from the control group.

The PRACTISS trial aims to improve treatment outcomes for patients with extremity STS by incorporating Liposomal Transcrocetin (L-TC) with Hypofractionated Radiotherapy (HFRT). L-TC is designed to enhance tumor oxygenation, addressing hypoxia-a significant factor contributing to radioresistance. By reoxygenating tumor cells, L-TC may improve radiosensitivity, increasing the efficacy of radiotherapy and leading to higher rates of pathological complete response (pCR) before surgery. Achieving a higher pCR is associated with better long-term outcomes and reduced recurrence rates. Additionally, the use of HFRT reduces the overall treatment schedule compared to conventional radiotherapy, minimizing the treatment burden for patients and potentially improving their quality of life while maintaining treatment effectiveness.

L-TC 300 mg QD, administered as intravenous infusion over 90 minutes, at a fixed dose of 300 mg daily before each HFRT fraction, for a total of 5 days corresponding to the planned five daily HFRT fractions. The intravenous infusion should start 120 minutes before each HFRT fraction. Radiotherapy is scheduled to coincide with the plasma peak, which occurs approximately 2 hours after the start of the infusion

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Localized or locally advanced soft tissue sarcoma of extremity proven by biopsy histological grade 2 and 3.
* Pathological expert proof-reading in reference centers
* HFRT and surgery planned (regardless the potential inclusion in this trial) as decided in a multidisciplinary tumor board, in reference centre (European Society for Medical Oncology (ESMO) guideline 2021)
* R0 surgery is feasible, in reference centers
* Pre-biopsy MRI available
* Performance status of 0-2 and life expectancy of at least 6 months

Exclusion Criteria:

* Patient who cannot undergo MRI
* Patients with localized or locally advanced soft tissue sarcoma of extremity proven by biopsy with histological grade 1
* Previous radiation in the area
* Woman who is pregnant or breastfeeding
* Soft tissue sarcoma developed in irradiated area.
* Patients with myxoid liposarcoma, embryonal or alveolar rhabdomyosarcoma, Ewing sarcoma, osteosarcoma, angiosarcoma, primitive neuroectodermal tumor, desmoid-type fibromatosis, or dermatofibrosarcoma protuberans
* Patient with metastatic disease, other concomitant cancer or history of cancer treated and controlled within the previous 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of the L-TC treatment in combination with preoperative hypofractionated radiotherapy (HFRT) | At surgery (Between 4 and 8 weeks after the end of radiotherapy)
  Pathological complete response rate (pCR): defined as the presence of < 10% residual malignant viable cells.

SECONDARY OUTCOMES:
Evaluation of the acute tolerance o f L-TC | Up to day 5 (every day during the treatment)
  Toxicities and biological analysis before each injection of L-TC and before surgery, described by type and grade, using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 classification
Evaluation of the late tolerance o f L-TC | Up to day 28 after the end of treatment.
  Toxicities and biological analysis before each injection of L-TC and before surgery, described by type and grade, using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 classification
Evaluation of the acute tolerance of radiotherapy | Up to day 5 (every day during the treatment)
  Global tolerance (radiotherapy toxicities (oedema, radiodermatitis, fibrosis, bone fracture) and laboratory abnormalities) at each physician consultation for radiotherapy and at follow-up, using the CTCAE v.5.0 classification
Evaluation of the late tolerance of radiotherapy | at 4 months after surgery, and at 12, 18, 24, 36 and 60 months
  Global tolerance (radiotherapy toxicities (oedema, radiodermatitis, fibrosis, bone fracture) and laboratory abnormalities) at each physician consultation for radiotherapy and at follow-up, using the CTCAE v.5.0 classification
Evaluation of tumour necrosis | At surgery (Between 4 and 8 weeks after the end of radiotherapy)
  Proportion of patient whom tumor has pathologic necrosis on histologic examination
Evaluation of the radiological response | at screening and before surgery
  Proportion of patients with a complete or partial radiological response (according to RECIST 1.1) evaluated on MRI
Proportion of patients with R0 resection | At surgery
  Number of patients with R0 resection on the number of enrolled patients
Evaluation of the Local Progression-Free Survival (L-PFS) | at 12, 24, 36 and 60 months.
  L-PFS will be defined as the length of time from the date of diagnostic by biopsy to the date of local relapse on MRI.
  L-PFS will be determined in median and rate
Evaluation of the Distant Progression-Free Survival (D-PFS) | at 12, 24, 36 and 60 months.
  D-PFS will be defined as the length of time from the date of diagnostic by biopsy to the date of distant relapse on scanner.
  D-PFS will be determined in median and rate
Evaluation of the Overall Survival (OS) | at 12, 24, 36 and 60 months
  OS will be defined as the length of time from the date of diagnostic by biopsy to the date of death, whatever the cause. Patients will be censored on the last news date.
  OS will be determined in median and rate
Evaluation of the Quality of Life (QoL) | at the inclusion (baseline) and every 4 months the two first years and then every 6 months the next three years
  Use of the European Organisation for Research and Treatment of Cancer (EORTC) 30-Item Core Quality of Life Questionnaire (QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle CHAMBRELANT, MD, Principal Investigator — Institut de cancérologie Strasbourg Europe; Georges NOEL, MD, PhD, Study Chair — Institut de cancérologie Strasbourg Europe
Locations (2):
- France (2):
  - CGFL, Dijon
  - ICANS, Strasbourg

IPD SHARING:
Plan to Share IPD: No